CLINICAL TRIAL: NCT04033133
Title: Cerebral Blood Flow in People With Multiple Sclerosis During Transcranial Direct Current Stimulation
Brief Title: Cerebral Blood Flow and tDCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Thorsten Rudroff, Assistant Professor, University of Iowa
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 201905826
Record Dates: First submitted 2019-07-23; First posted 2019-07-25 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; tDCS; Cerebral Blood Flow
MeSH Terms: conditions — Multiple Sclerosis | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: People with Multiple Sclerosis and healthy controls will receive tDCS at different intensities while in the PET scanner.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multiple Sclerosis (Experimental): People with MS get tDCS with different intensities.
  Interventions: Device: tDCS
- Healthy Subjects (Active Comparator): Healthy subjects get tDCS with different intensities.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — Subjects will get tDCS at intensities of 0, 1, 2, 3, and 4 mA.

SUMMARY:
With this study, the investigators will substantiate if regional cerebral blood flow (CBF) is affected by tDCS, assess the amount of CBF change in relation to different currents, and measure differences in regional CBF under stimulation reactivity between healthy subjects and people with Multiple Sclerosis (PwMS)using Water O-15 PET (Water Oxygen-15 Positron EmissionTomography) imaging. The objective is to investigate the changes in regional CBF after transcranial direct current stimulation (tDCS) at different intensities (1 mA, 2 mA, 3 mA, 4 mA) in healthy subjects and PwMS. The design is a cross-sectional proof of principle study in 10 healthy subjects and 10 PwMS.

Relative regional brain CBF (rCBF) will be analyzed semi-quantitatively using voxel-wise and region of interest-based approaches. Changes in CBF associated with tDCS-application will be calculated with a general linear model in a ramp function of the task-specific rCBF, according to previous work in our group using a glucose analogue. Exploratory statistical testing will be done using a paired samples t-test between task and rest conditions and unpaired t-tests between PwMS and healthy controls at the same intensities.

With this study the investigators will be able to dose-dependently measure real-time rCBF changes after non-invasively stimulating the superficial parts of the dorsolateral prefrontal cortex (DLPFC), a commonly used target in therapeutic tDCS applications. This will provide further insight into whether tDCS is capable of inducing changes in rCBF.

DETAILED DESCRIPTION:
Aim 1: To determine the effects of different stimulation intensities on relative cerebral blood flow (rCBF).

Currently, researchers use tDCS as an interventional modality to modulate the excitability of the brain, with measureable changes in both motor evoked potentials and physical performances. However, because of the relatively large size of most electrodes, and the electrodynamics of the brain, it still remains unclear what specific brain structures are being stimulated and how the mechanics of stimulation (e.g., stimulation penetration and areas affected outside of target area) change with different intensities. The investigators hypothesize that regional CBF at the DLPFC (target area) will increase in a dose-dependent way with greater stimulation intensity. Furthermore, it is hypothesized that the areas surrounding the DLPFC will be increasingly affected by higher stimulation intensities.

Aim 2: To contrast the effects of transcranial direct current stimulation on relative cerebral blood flow between healthy subjects and people with Multiple Sclerosis.

PwMS typically present with glucose hypometabolism compared to their healthy peers and because CBF and glucose metabolism are highly coupled, a similar trend in CBF may be expected. Additionally, tDCS has been shown to be effective at increasing cortical excitability and glucose metabolism in both populations. However, what still remains uncertain is if PwMS and healthy subjects experience the same amount of increased activity for the same stimulation intensity. The investigators hypothesize that PwMS will experience a greater increase in rCBF at the DLPFC and surrounding areas than healthy controls for the same stimulation intensity.

Aim 3: To extend our understanding of the safety and efficacy of transcranial direct current stimulation at higher current intensities for healthy subjects and people with Multiple Sclerosis.

Despite some work on the feasibility and safety of performing tDCS at intensities > 2 mA (i.e., up to 4 mA), the convention for most tDCS studies is to use intensities less than or equal to 2 mA. This has been sufficient to illicit measurable effects in both excitability and performance outcomes. However, the potential benefits of increasing intensity to either enhance the effects of a given stimulation protocol (e.g., time or magnitude) or to potentially access deeper brain areas justifies further exploration of current intensities > 2 mA. It is also important to add to the safety protocol of higher intensities in healthy and clinical (e.g., PwMS) subjects. The investigators hypothesize that higher intensities (i.e., > 2 mA) will be well tolerated by both healthy subjects and PwMS. Additionally, the investigators hypothesize no serious adverse effects from higher stimulation intensities. The existing side-effects of tDCS at intensities less than or equal to 2 mA include low-grade occurrences of tingling, itching, and burning sensation at the electrode sites; a few subjects have reported short-lived (< 5 min) headaches. In a study testing the safety of higher intensities similar to those proposed here, these same side-effects were observed in 50% of the subjects. This rate of occurrence is slightly higher than studies using less than or equal to 2 mA, but the magnitudes of the negative effects were still well within safely tolerable limits and were all transient in nature.

I.6 Background and significance and/or Preliminary studies related to this project.

(do not indicate "see protocol") Transcranial direct current stimulation (tDCS) is a non-invasive and well-tolerated brain stimulation technique (1-4) that can modulate the cortical excitability of targeted brain regions (5) as well as cerebral blood flow (6) in a polarity-dependent manner.

Models of tDCS current flow (7,8) and findings from studies in which human functional magnetic resonance Imaging (fMRI) has been used to measure brain activity (9-11) suggest that tDCS can alter processing across large areas of the cortex. In this sense, the effects of tDCS are likely to be relatively broad. Thus, while the neural changes induced by tDCS are concentrated around regions of cortex closest to the electrodes (12), broader networks of functionally-connected regions may also be recruited (9,10,13,14). Furthermore, no systematic investigation has been done to determine the most efficacious current intensity for PwMS.

There is empirical evidence that tDCS with current intensity between 1 and 2 mA for 20-40 minutes for either single or multiple sessions can safely and effectively be administered to PwMS (15-20). Although tDCS with current intensities > 2 mA are considered safe 21, no studies have investigated how brain activity is affected during tDCS at intensities > 2 mA. Although the safety of higher intensity tDCS in PwMS may be initially assumed from previous work using subjects who have experienced a stroke (21), it has also been suggested that more studies on the safety of higher intensity stimulation in other populations are needed in order to exercise due diligence before widely prescribing intensities greater than the present convention (22).

The cerebral activation in PwMS has been investigated with [15O] water and with [15O] O2 PET (indexes oxygen metabolism)(23). Widespread reductions in cerebral blood flow and oxygen metabolism in both gray and white mater have been reported in PwMS (24). Furthermore, these studies indicate that the degree of oxygen metabolism reduction correlated with worse cognitive performance and expanded disability status scale (EDSS), and that the degree of cerebral oxygen hypometabolism was associated with the number of relapses (25).

A close coupling of perfusion and metabolism is assumed, reflecting oxidative phosphorylation of glucose as the predominant source of energy production. Consequently, CBF is often considered as an indirect measure of neuronal function and integrity (26). This is supported by the significant association of metabolism with regional CBF (rCBF) across different brain regions (27,28), and with global CBF (gCBF) across varying states of consciousness (29).

With this study, the investigators will be able to substantiate if rCBF is affected by tDCS, assess the amount of signal change in relation to different currents, and measure differences in CBF distribution under stimulation reactivity between healthy subjects and PwMS. The objective is to investigate the changes in rCBF after transcranial direct current stimulation at different intensities (1 mA, 2 mA, 3 mA, 4 mA) in healthy subjects and PwMS. The design is a cross-sectional proof of principle study in 10 healthy subjects and 10 PwMS.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of multiple sclerosis by a neurologist
* No change in MS-specific medication (disease modification drugs) in the last three months
* Healthy enough to complete the protocol based on information obtained from a clinical exam and past medical history.
* An expanded disability status scale (EDSS) below 5.5
* Comprehension of the protocol as indicated by an ability to respond to questions about the study after reading the consent form.
* Able to use and be contacted by telephone
* Able to speak, read, and understand English, and complete a questionnaire in English
* Body mass index <30 kg/m2

Exclusion Criteria:

* A relapse of disease symptoms in the last three months
* History / presence of secondary conditions such as seizure disorders (or on medications known to lower seizure threshold), hydrocephalus, diabetes mellitus, or claustrophobia
* Alcohol dependence or abuse (>2 drinks/day), or present history (last six months) of drug abuse
* History of significant traumatic brain injury or hydrocephalus
* Currently pregnant
* Recent hospitalization (within the last 3 months) or enforced bed rest/sedentary state
* Claustrophobia

A subject will be excluded if he/she has a contraindication to Magnetic Resonance scanning, e.g., implanted metal clips or wires, which may concentrate radiofrequency fields or cause tissue damage from twisting in a magnetic field.

Examples include:

* Aneurysm clip
* Implanted neural stimulator
* Implanted cardiac pacemaker or autodefibrillator
* Cochlear implant
* Ocular foreign body (e.g., metal shavings)
* Any implanted device (pumps, infusion devices, etc.)
* Shrapnel injuries

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Cerebral Blood Flow | Through study completion, an average of 1 year
  Cerebral Blood flow will be measured while subjects undergo tDCS at different intensities in the PET scanner.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Health and Human Physiology, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No